CLINICAL TRIAL: NCT03256266
Title: Establishment of Small Intestinal Human Organoids to Check the Influence of Nutrient Antigens or Therapeutic Agents
Brief Title: Effect of Antigens or Therapeutic Agents on in Vitro Human Intestinal Organoids
Status: Active, not recruiting | Type: Observational
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Other Study IDs: intestinal organoids
Record Dates: First submitted 2017-05-31; First posted 2017-08-22 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Intestine Disease
MeSH Terms: conditions — Intestinal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- healthy controls: healthy controls
- patients with allergy: patients with Food intolerances or Food allergy
- gastrointestinal disorders: patients with inflammatory bowel disease, irritable bowel disease, gluten sensitivity, short bowel syndrome

SUMMARY:
The study evaluates the effect of nutrient antigens or therapeutic agents on human small intestinal organoids.

DETAILED DESCRIPTION:
Small intestinal biopsies will be taken to establish human intestinal organoids in vitro. The organoids will be propagated and various antigens will be checked for their effects on proliferation, production of inflammatory components or signal cascade.

ELIGIBILITY:
Inclusion Criteria:

* patients with gastrointestinal disorders and therapeutical indication of gastroduodenoscopy or coloscopy
* healthy controls for preventive medical check-up

Exclusion Criteria:

* pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: -Patients with patients with Food intolerances, Food allergy, intestinal disorders, glutensensitivity, healthy controls who underwent a gastroduodenoscopy or coloscopy for therapeutical intervention or screening
Sampling Method: Non-Probability Sample
Enrollment: 375 (Estimated)
Dates: Start 2017-04-01 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Determination of proliferation, apoptosis, histology, and cytokine Expression before and after Antigen provocation of organoids with gluten peptides, nutritional Antigens, Glucagon like peptide antagonist, or Tumor nekrose factor antagonists | baseline vs 24h vs 48h vs 72h
  Determination of effects on organoids after antigen Stimulation with ELISA, histochemistry, RNA or proteome analysis

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Medicine 1, Hector Center for Nutrition, Exercise and Sports, Friedrich-Alexander-University Erlangen-Nuremberg, Erlangen, Germany

IPD SHARING:
Plan to Share IPD: No